CLINICAL TRIAL: NCT04068337
Title: Freestyle Prosthesis for Aortic Root-replacement With and Without Hemiarch Replacement in Various Pathologies: A Retrospective Analysis
Brief Title: Freestyle Prosthesis for Aortic Root-replacement With and Without Hemiarch Replacement
Status: Completed | Type: Observational
Sponsor: Triemli Hospital (Other)
Responsible Party: Principal Investigator, Alicja Zientara, resident for cardiac surgery, Triemli Hospital
Other Study IDs: BASEC-Nr. 2018-01227
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Aortic Aneurysm; Aortic Dissection; Endocarditis; Root Abscess; Valve Heart Disease
Keywords: hemiarch replacement; cardiopulmonary bypass; cannulation technique; selective cerebral perfusion
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection; Endocarditis; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemiarch: Patients with Freestyle aortic root implantation receiving a hemiarch replacement by open anastomosis technique with axillary cannulation and antegrade cerebral perfusion
  Interventions: Procedure: Aortic root replacement with Freestyle biological prosthesis with and without hemiarch replacement
- Non-Hemiarch: Patients with Freestyle aortic root implantation without hemiarch replacement with normal systemic perfusion
  Interventions: Procedure: Aortic root replacement with Freestyle biological prosthesis with and without hemiarch replacement

INTERVENTIONS:
Procedure: Aortic root replacement with Freestyle biological prosthesis with and without hemiarch replacement — Aortic root replacement with Freestyle biological prosthesis. Some patients receive additional hemiarch replacement performing an open anastomosis to the aortic arch under antegrade cerebral perfusion through axillary artery. Comparison with patients, who were cannulated and perfused systemically

SUMMARY:
The Freestyle® prosthesis (Medtronic plc, Dublin, Ireland) is a biological, porcine aortic root implanted in various combinations and techniques since the 1990s. The main indication for the choice of this prosthesis is a combined pathology with degenerated aortic valve and additional dilatation of the root often involving the ascending aorta.

The Freestyle® prosthesis is also used in cases of dissection of the ascending aorta with the involvement of the aortic valve, which opens the debate on how far the ascending aorta should be replaced for a sustainable solution with calculable low periprocedural risk. Considering a lower intraoperative risk in the life-threatening situation, an extended resection of the aorta can be avoided and only the aortic root replaced with a piece of ascending aorta. On the contrary, focusing on improved long-term outcome, the technique of total arch replacement in aortic dissection was developed in emergency situations with acceptable results, which, however, were often reproducible only in large, experienced centers.

Apart from the abovementioned options, the technique of proximal arch replacement can provide a tension-free anastomosis. The intention of hemiarch replacement is the attachment of the prosthesis to an aneurysm-free portion of the aortic arch helping to protect against further anastomotic aneurysms and spare the patient complex reoperation or interventional procedures in the future. As a possible drawback of the technique, especially in emergency situations, the potentially prolonged duration of surgery and the need of selective brain perfusion via axillary or carotid artery are discussed increasing the risk of stroke and further major events, which could not be reflected in current literature. However, there is still no convincing evidence of a long-term benefit in terms of re-operation and survival after hemiarch replacement.

The aim of this retrospective analysis was to assess the mid-term outcome of the biological Freestyle® prosthesis in combination with operations on the ascending aorta and the aortic arch with regard to prosthetic performance, reoperations, stroke and death.

ELIGIBILITY:
Inclusion Criteria:

* all patients after implantation of a biological Medtronic Freestyle root prosthesis in the time frame from November 2007 till April 2017
* elective, urgent and emergency operations on ascending aneurysms, aortic dissections, endocarditis and aortic root pathologies
* combination of other procedures (coronary artery bypass grafting, operations on mitral and tricuspid valve, ablations)

Exclusion Criteria:

* refused patient consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From September 2007 till March 2017, we performed 278 aortic root replacements with the Freestyle prosthesis at a single centre in Switzerland. Two groups were identified based on the additional replacement of the hemiarch resulting in 119 patients (HA) and 159 patients without an additional hemiarch replacement (non-HA). Patients with additional valve and coronary artery procedures were included as well. Out of the non-HA group, 7 patients were cannulated through the femoral artery and excluded for further analysis.
Sampling Method: Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days after initial operation
  In-hospital mortality
Major and minor in-hospital complications | 30 days after initial operation
  stroke, myocardial infarction, re-operation, pacemaker implantation
Valve performance | earliest to longest follow up (longest follow up period of 10 years)
  Mean valve gradient of the implanted root prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Alicja Zientara, MD, Principal Investigator — Triemli Hospital
Locations (1):
- Triemli Hospital, Zurich, Switzerland